CLINICAL TRIAL: NCT05815043
Title: Effects of Sodium Intake on Arterial Stiffness in Black Adults
Brief Title: Effects of Sodium Intake on Arterial Stiffness in Black Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 8663
Record Dates: First submitted 2023-02-22; First posted 2023-04-18 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Sodium Intake; Arterial Stiffness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low- and high-sodium intake (Experimental): Participants will consume two different quantities of sodium per day for 3 days each.
  Interventions: Behavioral: Low-sodium intake; Dietary Supplement: High-sodium intake

INTERVENTIONS:
Behavioral: Low-sodium intake — Participants will consume less than or equal to 720 milligrams of sodium per day for 3 days.
Dietary Supplement: High-sodium intake — Participants will supplement their existing diets with 10 salt tablets daily for 3 days.

SUMMARY:
The purpose of this study is to explore the influence of sodium intake on arterial stiffness in African American/Black adults.

ELIGIBILITY:
Inclusion Criteria:

* African American or Black
* Male or Female

Exclusion Criteria:

* pregnancy or within 60 days postpartum
* having taken blood pressure (including diuretics beta-blockers, ACE inhibitors, angiotensin receptor blockers, and calcium channel blockers) or statin medications within the past 3 months
* infection (viral or other) within the past 4 weeks
* having adrenal or endocrine tumors (these could impact BP)
* renal disease defined as a glomerular filtration rate (GFR) of less than 60
* prior myocardial infarction
* known coronary heart disease
* personal history of stroke
* heart failure
* cardiac arrhythmias
* recent chest pain or dyspnea
* current insulin dependence
* currently undergoing chemotherapy or radiation
* identifying as transgender (the focus of this trial is biological sex)
* seated systolic or diastolic blood pressure of more than 149 mm Hg or 99 mm Hg, respectively

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Cardio-ankle vascular index | This measurement will take approximately 1 minute and will be completed twice.
  Cardio-ankle vascular index will be assessed using simultaneous arm and ankle blood pressures, EKG, and phonocardiography
Ambulatory blood pressure | This measurement will take approximately 24 hours and will be obtained from the date of enrollment until the date of completion of the study up to 10 days after enrollment.
  24-hour ambulatory blood pressure monitoring will be completed on day 3 of each dietary condition.

SECONDARY OUTCOMES:
Renal sodium excretion | This measurement will be obtained from the date of enrollment until the date of completion of the study up to 10 days after enrollment.
  24-hour urine samples will be analyzed for sodium concentrations and sodium excretion will be determined.

OTHER OUTCOMES:
Hematocrit | This measurement will be obtained from the date of enrollment until the date of completion of the study up to 10 days after enrollment.
  Hematocrit will be determined from whole blood samples after each 3-day dietary condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas State University, San Marcos, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided